CLINICAL TRIAL: NCT00258258
Title: An Open Label Dose Escalation Study of Intravenous Paricalcitol (ZEMPLAR™) [19-NOR-1 ALPHA, 25 - (OH)D] With Zoledronic Acid (Zometa™) in Patients With Multiple Myeloma
Brief Title: Paricalcitol and Zoledronate in Treating Patients With Relapsed or Refractory Multiple Myeloma or Other Plasma Cell Disorders
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn due to low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: I 38504; RPCI-I-38504; NOVARTIS-RPCI-I-38504; ABBOTT-RPCI-I-38504
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — paricalcitol; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: paricalcitol
Drug: zoledronic acid

SUMMARY:
RATIONALE: Paricalcitol may cause multiple myeloma cells to look more like normal cells, and to grow and spread more slowly. Paricalcitol may also stop the growth of the cancer cells by blocking blood flow to the cancer. Zoledronate may delay or prevent bone metastases in patients with multiple myeloma. Giving paricalcitol together with zoledronate may be an effective treatment for multiple myeloma or other plasma cell disorders.

PURPOSE: This clinical trial is studying the side effects and best dose of paricalcitol when given with zoledronate in treating patients with relapsed or refractory multiple myeloma or other plasma cell disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of paricalcitol when used with zoledronate in patients with relapsed or refractory multiple myeloma or other plasma cell disorders.

Secondary

* Determine the toxic effects of this regimen in these patients.
* Determine the antimyeloma activity of paricalcitol in patients treated with this regimen.

OUTLINE: This is an open-label, dose-escalation study of paricalcitol.

Patients receive paricalcitol IV over 15 minutes on days 1, 8, and 15 and zoledronate IV over 15 minutes on day 22. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of paricalcitol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of relapsed or refractory multiple myeloma (MM) or other plasma cell disorder (PCD)

  * At least one previous treatment for MM or PCD required

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* At least 3 months

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Calcium ≤ 10.5 mg/dL
* No renal stone formation within the past 5 years for patients who have had curative therapy for a condition associated with the risk of stones (e.g., hyperparathyroidism, bladder dysfunction, obstructive uropathy) OR had a single episode of confirmed urolithiasis
* No calculi in urinary tract confirmed by renal ultrasonography, kidney, ureter, and bladder (KUB) x-ray, or other imaging modality

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No uncontrolled cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during study and for 3 months after study completion
* No osteonecrosis of the jaw
* No history of allergic reaction attributed to compounds of similar chemical or biological composition of calcitriol, paricalcitol, or zoledronate
* No uncontrolled intercurrent illness that would preclude study compliance
* No ongoing or active infection
* No psychiatric illness or social situation that may preclude study compliance

PRIOR CONCURRENT THERAPY:

Chemotherapy

* More than 4 weeks since prior chemotherapy

Endocrine

* More than 4 weeks since prior high-dose steroids

Other

* No other concurrent investigational agents or therapies for multiple myeloma or plasma cell disorders
* No concurrent digoxin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-08; Primary Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asher A. Chanan-Khan, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States